CLINICAL TRIAL: NCT05753683
Title: GODDESS (Gathering Online for Dialogue and Discussion to Enhance Social Support): Engaging Young African American Women in a Virtual Group App to Address Alcohol Misuse, Sexual Risk, and Pre-exposure Prophylaxis (PrEP) in North Carolina (NC)
Brief Title: Gathering Online for Dialogue and Discussion to Enhance Social Support
Acronym: GODDESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Felicia A. Browne, ScD, MPH, Senior Research Social Epidemiologist, RTI International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0218271; R01AA030452 (NIH)
Record Dates: First submitted 2023-01-06; First posted 2023-03-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Misuse; HIV; Sexually Transmitted Infections; Pre-exposure Prophylaxis
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard: mHealth-Women's CoOp (Active Comparator): Participants assigned to receive an evidence-based mHealth alcohol and other drug use and sexual risk reduction intervention for young African American women. The app will be installed on each participant's smartphone by study staff after randomization.
  Interventions: Behavioral: mHealth-Women's CoOp
- Enhanced: mHealth-Women's CoOp+Group (Experimental): Participants assigned to receive an evidence-based mHealth alcohol and other drug use and sexual risk reduction intervention for young African American women, in addition to a virtual peer group component. The app with a link to the virtual group will be installed on each participant's smartphone by study staff after randomization.
  Interventions: Behavioral: mHealth-Women's CoOp; Behavioral: Virtual Group

INTERVENTIONS:
Behavioral: mHealth-Women's CoOp — The mHealth-Women's CoOp, was developed and tested in a previous randomized trial, is a human immunodeficiency virus (HIV) risk-reduction intervention that addresses the intersection of substance use, sexual risk and violence through education, skills-building, and role-play and rehearsal via a mobile app. The mHealth-Women's CoOp app is also used to help participants monitor progress toward their goals throughout the study period. Specifically, the app is programmed to prompt the user, to visit the app and participate in several activities, including health and behavior check-in and revisiting aspects of the mHealth-Women's CoOp educational content to sustain risk reduction.
Behavioral: Virtual Group — The enhanced online group component will be available to be accessed using the mHealth-Women's CoOp platform for participants in the enhanced arm. The purpose of this component is to allow for young women who use alcohol to interact with young women like them and also discuss issues related to substance use and sexual risk-taking via a guided conversation to allow for motivational and informational support. The virtual group component will include online live discussions moderated and monitored by a trained online facilitator.
  Arms: Enhanced: mHealth-Women's CoOp+Group

SUMMARY:
The goal of this trial is to test a modified mobile health intervention (with a group component) relative to a mobile health intervention in a two-arm randomized trial with 500 young African American women who are human immunodeficiency virus (HIV)-negative and who misuse alcohol.

The expected outcomes are to: (1) determine the efficacy of the virtual group component in reducing alcohol use and sexual risk and increasing pre-exposure prophylaxis (PrEP) utilization; and (2) understand selected outcomes for implementation.

Participants will be randomized to receive either the mHealth app or the mHealth app plus the group component, and followed up at 3- and 6-months post-enrollment.

DETAILED DESCRIPTION:
A total of 500 participants who are human immunodeficiency virus (HIV)-negative who engage in heavy alcohol use will be enrolled and referred to their local health departments for pre-exposure prophylaxis (PrEP). Primary biobehavioral outcomes assessed will include reduced alcohol use (self-reported and biological, including phosphatidylethanol [PEth]), increased PrEP uptake (self-reported and biological), and reduced sexual risk (self-reported condomless sex and impaired sex and biological testing for HIV) at 3- and 6-month follow-up.

ELIGIBILITY:
Selected Inclusion Criteria:

* identify as Black/African American
* identify as female
* be between 18 and 30 years old
* recent substance use
* HIV negative and not currently on PrEP
* have an Android or iOS-based smartphone

Selected Exclusion Criteria:

* test positive for HIV
* participated in the previous study activities of the current study or previous related studies

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Identify as female
Enrollment: 500 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Alcohol (Biological) | Baseline
  Recent alcohol (last 10 days) use will be measured by the presence of ethyl glucuronide (EtG), a breakdown product of ethanol, using an ethyl glucuronide (EtG) urine test. The One Step Ethyl Glucuronide (EtG) Test Dip Card is a lateral flow chromatographic immunoassay. Each test has a control line region to serve as a procedural control and a test line region; results with only a line in the control region and without a line in the test region are classified as positive. Urine EtG ≥300 ng/mL indicates a positive result.
Alcohol (Biological) | 3-month
  Recent alcohol (last 10 days) use will be measured by the presence of ethyl glucuronide (EtG), a breakdown product of ethanol, using an ethyl glucuronide (EtG) urine test. The One Step Ethyl Glucuronide (EtG) Test Dip Card is a lateral flow chromatographic immunoassay. Each test has a control line region to serve as a procedural control and a test line region; results with only a line in the control region and without a line in the test region are classified as positive. Urine EtG ≥300 ng/mL indicates a positive result.
Alcohol (Biological) | 6-month
  Recent alcohol (last 10 days) use will be measured by the presence of ethyl glucuronide (EtG), a breakdown product of ethanol, using an ethyl glucuronide (EtG) urine test. The One Step Ethyl Glucuronide (EtG) Test Dip Card is a lateral flow chromatographic immunoassay. Each test has a control line region to serve as a procedural control and a test line region; results with only a line in the control region and without a line in the test region are classified as positive. Urine EtG ≥300 ng/mL indicates a positive result.
Alcohol (Biological) | Baseline
  Phosphatidylethanol (PEth) in dried blood spots (DBS) with concentration equal to or greater than 8 ng/mL is an indication of alcohol exposure in the last 2-4 weeks (approximately). Higher concentrations of PEth indicates higher recent alcohol consumption.
Alcohol (Biological) | 3-month
  Phosphatidylethanol (PEth) in dried blood spots (DBS) with concentration equal to or greater than 8 ng/mL is an indication of alcohol exposure in the last 2-4 weeks (approximately). Higher concentrations of PEth indicates higher recent alcohol consumption.
Alcohol (Biological) | 6-month
  Phosphatidylethanol (PEth) in dried blood spots (DBS) with concentration equal to or greater than 8 ng/mL is an indication of alcohol exposure in the last 2-4 weeks (approximately). Higher concentrations of PEth indicates higher recent alcohol consumption.
Alcohol (Self-Reported) | Baseline
  Revised Risk Behavior Assessment (RRBA): Volume (grams of ethanol, accounting for different standard drink size), frequency of use, frequency of binge, heavy episodic drinking (4+ drinks/day).
Alcohol (Self-Reported) | 3-month
  Revised Risk Behavior Assessment (RRBA): Volume (grams of ethanol, accounting for different standard drink size), frequency of use, frequency of binge, heavy episodic drinking (4+ drinks/day).
Alcohol (Self-Reported) | 6-month
  Revised Risk Behavior Assessment (RRBA): Volume (grams of ethanol, accounting for different standard drink size), frequency of use, frequency of binge, heavy episodic drinking (4+ drinks/day).
Alcohol (Self-Reported) | Baseline
  World Health Organization's Alcohol, Smoking & Substance Use Involvement Scale (ASSIST) assesses risk for alcohol consumption problems via 8 items. Scores range from 0 to 39, and this score indicates level of risk for alcohol consumption problems. Scores from 0 to 10 indicate lower risk for alcohol problems, scores from 11 to 26 indicate moderate risk, and scores from 27 to 39 indicate high risk.
Alcohol (Self-Reported) | 3-month
  World Health Organization's Alcohol, Smoking & Substance Use Involvement Scale (ASSIST) assesses risk for alcohol consumption problems via 8 items. Scores range from 0 to 39, and this score indicates level of risk for alcohol consumption problems. Scores from 0 to 10 indicate lower risk for alcohol problems, scores from 11 to 26 indicate moderate risk, and scores from 27 to 39 indicate high risk.
Alcohol (Self-Reported) | 6-month
  World Health Organization's Alcohol, Smoking & Substance Use Involvement Scale (ASSIST) assesses risk for alcohol consumption problems via 8 items. Scores range from 0 to 39, and this score indicates level of risk for alcohol consumption problems. Scores from 0 to 10 indicate lower risk for alcohol problems, scores from 11 to 26 indicate moderate risk, and scores from 27 to 39 indicate high risk.
Sexual Risk: HIV (Biological) | Baseline
  Number of participants living with HIV as assessed by OraQuick® ADVANCE Rapid HIV-1/2 Antibody Test with oral fluid, with an approximate 99.3% sensitivity & 99.8% specificity, which detects antibodies to HIV-1 and HIV-2.
Sexual Risk: HIV (Biological) | 6-month
  Number of participants living with HIV as assessed by OraQuick® ADVANCE Rapid HIV-1/2 Antibody Test with oral fluid, with an approximate 99.3% sensitivity & 99.8% specificity, which detects antibodies to HIV-1 and HIV-2.
Sexual Risk (Self-reported) | Baseline
  Revised Risk Behavior Assessment (RRBA): Condomless vaginal or anal sex, impaired sex (AOD use prior to or during sex), casual partners, sex trading, & concurrent partners (≥2 partners), other contraceptive use, & perception of risk, HIV, recent STIs
Sexual Risk (Self-reported) | 3-month
  Revised Risk Behavior Assessment (RRBA): Condomless vaginal or anal sex, impaired sex (AOD use prior to or during sex), casual partners, sex trading, & concurrent partners (≥2 partners), other contraceptive use, & perception of risk, HIV, recent STIs
Sexual Risk (Self-reported) | 6-month
  Revised Risk Behavior Assessment (RRBA): Condomless vaginal or anal sex, impaired sex (AOD use prior to or during sex), casual partners, sex trading, & concurrent partners (≥2 partners), other contraceptive use, & perception of risk, HIV, recent STIs
PrEP Utilization (Biological) | 3-month
  Dried blood spot (DBS) samples will be analyzed by quantification of drug concentrations by liquid chromatography-tandem mass spectrometry (LC-MS/MS) technology using assays validated at the study laboratory.
PrEP Utilization (Biological) | 6-month
  Dried blood spot (DBS) samples will be analyzed by quantification of drug concentrations by liquid chromatography-tandem mass spectrometry (LC-MS/MS) technology using assays validated at the study laboratory.
PrEP Utilization (Self-Reported) | Baseline
  Revised Risk Behavior Assessment (RRBA): Self-reported past 30-day use, missed doses, and patterns of use
PrEP Utilization (Self-Reported) | 3-month
  Revised Risk Behavior Assessment (RRBA): Self-reported past 30-day use, missed doses, and patterns of use
PrEP Utilization (Self-Reported) | 6-month
  Revised Risk Behavior Assessment (RRBA): Self-reported past 30-day use, missed doses, and patterns of use

SECONDARY OUTCOMES:
Drug Use (Biological) | Baseline
  Easy@Home Multi-Drug Screen Test: Rapid urine-based drug screen to detect metabolites of recent drug use (>99% correlation to gas chromatography at 95% confidence level) 10-panel-amphetamine, benzodiazepines, barbiturates, cocaine, opiates, methamphetamine, ecstasy, methadone, phencyclidine, and marijuana. Each test has a control line region to serve as a procedural control and a test line region; results with only a line in the control region and without a line in the test region are classified as positive. Concentrations at or above the following cutoff concentrations indicate a positive result for the following substances: amphetamine (1000 ng/mL), benzodiazepines (300 ng/mL), barbiturates (300 ng/mL), cocaine (300 ng/mL), opiates (2000 ng/mL), methamphetamine (1000 ng/mL), ecstasy (500 ng/mL), methadone (300 ng/mL), phencyclidine (25 ng/mL), marijuana (50 ng/mL).
Drug Use (Biological) | 3-month
  Easy@Home Multi-Drug Screen Test: Rapid urine-based drug screen to detect metabolites of recent drug use (>99% correlation to gas chromatography at 95% confidence level) 10-panel-amphetamine, benzodiazepines, barbiturates, cocaine, opiates, methamphetamine, ecstasy, methadone, phencyclidine, and marijuana. Each test has a control line region to serve as a procedural control and a test line region; results with only a line in the control region and without a line in the test region are classified as positive. Concentrations at or above the following cutoff concentrations indicate a positive result for the following substances: amphetamine (1000 ng/mL), benzodiazepines (300 ng/mL), barbiturates (300 ng/mL), cocaine (300 ng/mL), opiates (2000 ng/mL), methamphetamine (1000 ng/mL), ecstasy (500 ng/mL), methadone (300 ng/mL), phencyclidine (25 ng/mL), marijuana (50 ng/mL).
Drug Use (Biological) | 6-month
  Easy@Home Multi-Drug Screen Test: Rapid urine-based drug screen to detect metabolites of recent drug use (>99% correlation to gas chromatography at 95% confidence level) 10-panel-amphetamine, benzodiazepines, barbiturates, cocaine, opiates, methamphetamine, ecstasy, methadone, phencyclidine, and marijuana. Each test has a control line region to serve as a procedural control and a test line region; results with only a line in the control region and without a line in the test region are classified as positive. Concentrations at or above the following cutoff concentrations indicate a positive result for the following substances: amphetamine (1000 ng/mL), benzodiazepines (300 ng/mL), barbiturates (300 ng/mL), cocaine (300 ng/mL), opiates (2000 ng/mL), methamphetamine (1000 ng/mL), ecstasy (500 ng/mL), methadone (300 ng/mL), phencyclidine (25 ng/mL), marijuana (50 ng/mL).
Drug Use (Self-Reported) | Baseline
  The World Health Organization's Alcohol, Smoking & Substance Use Involvement Scale (ASSIST) assesses risk for problems with drugs-such as marijuana, cocaine, amphetamine, and opioids-via 8 items. Scores range from 0 to 39, and this score indicates level of risk for drug use problems. Scores from 0 to 3 indicate lower risk for drug use problems, scores from 4 to 26 indicate moderate risk, and scores from 27 to 39 indicate high risk.
Drug Use (Self-Reported) | 3-month
  The World Health Organization's Alcohol, Smoking & Substance Use Involvement Scale (ASSIST) assesses risk for problems with drugs-such as marijuana, cocaine, amphetamine, and opioids-via 8 items. Scores range from 0 to 39, and this score indicates level of risk for drug use problems. Scores from 0 to 3 indicate lower risk for drug use problems, scores from 4 to 26 indicate moderate risk, and scores from 27 to 39 indicate high risk.
Drug Use (Self-Reported) | 6-month
  The World Health Organization's Alcohol, Smoking & Substance Use Involvement Scale (ASSIST) assesses risk for problems with drugs-such as marijuana, cocaine, amphetamine, and opioids-via 8 items. Scores range from 0 to 39, and this score indicates level of risk for drug use problems. Scores from 0 to 3 indicate lower risk for drug use problems, scores from 4 to 26 indicate moderate risk, and scores from 27 to 39 indicate high risk.
Perceived social support | Baseline
  Multidimensional Scale of Perceived Social Support assesses perceived social support Multidimensional Scale of Perceived Social Support assesses perceived social support from family, friends, and others across a 12-item scale. Each item uses a 7-point scale (1 = very strongly disagree, 7 = very strongly agree). Items are summed and the total score is divided by the number of items. Scores range from 0 to 7. Higher scores indicate higher levels of social support.
Perceived social support | 3-month
  Multidimensional Scale of Perceived Social Support assesses perceived social support from family, friends, and others across a 12-item scale. Each item uses a 7-point scale (1 = very strongly disagree, 7 = very strongly agree). Items are summed and the total score is divided by the number of items. Scores range from 0 to 7. Higher scores indicate higher levels of social support.
Perceived social support | 6-month
  Multidimensional Scale of Perceived Social Support assesses perceived social support from family, friends, and others across a 12-item scale. Each item uses a 7-point scale (1 = very strongly disagree, 7 = very strongly agree). Items are summed and the total score is divided by the number of items. Scores range from 0 to 7. Higher scores indicate higher levels of social support.
Violence | Baseline
  Adaptation of the World Health Organization (WHO) violence scale: Self-reported occurrence of emotional, physical, and sexual violence with an additional financial abuse query, all combined into a 16-item scale. Each item uses a 3-point response scale (1 = Never, 2 = Sometimes, 3 = Frequently). Items are summed, and scores range from 16 to 48. Higher scores indicate more frequent occurrences of violence.
Violence | 3-month
  Adaptation of the World Health Organization (WHO) violence scale: Self-reported occurrence of emotional, physical, and sexual violence with an additional financial abuse query, all combined into a 16-item scale. Each item uses a 3-point response scale (1 = Never, 2 = Sometimes, 3 = Frequently). Items are summed, and scores range from 16 to 48. Higher scores indicate more frequent occurrences of violence.
Violence | 6-month
  Adaptation of the World Health Organization (WHO) violence scale: Self-reported occurrence of emotional, physical, and sexual violence with an additional financial abuse query, all combined into a 16-item scale. Each item uses a 3-point response scale (1 = Never, 2 = Sometimes, 3 = Frequently). Items are summed, and scores range from 16 to 48. Higher scores indicate more frequent occurrences of violence.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia A Browne, ScD, MPH, Principal Investigator — RTI International
Locations (1):
- RTI International, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] van der Drift IM, Browne FA, Nyamaizi AM, Wechsberg WM. "A lot of the answers come from within you as well": benefits and limitations to utilizing and adapting a virtual platform to enhance social interaction and group learning. BMC Digit Health. 2025;3(1):64. doi: 10.1186/s44247-025-00204-1. Epub 2025 Sep 22. PMID 40989241